CLINICAL TRIAL: NCT01467687
Title: Comparative, Randomized, Single-Dose, 2-way Crossover Bioavailability Study of Synerx Pharma and Verelan PM 300 mg Verapamil HCl Extended Release Capsules Controlled-Onset in Healthy Aduly Volunteers Under Fed Conditions
Brief Title: Comparative Bioavailability Study of Synerx and Verelan PM 300 mg Verapamil HCl ER Capsules Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Synerx Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AA32724
Record Dates: First submitted 2011-10-31; First posted 2011-11-09 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-11

CONDITIONS: Healthy
MeSH Terms: interventions — Verapamil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 300 mg capsule of Verelan PM or 300 mg verapamil controlled release capsule given orally with food as a single dose with blood collected at 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 14, 16, 24, 30, 36, 48, 60 and 72 hours.
  Interventions: Drug: verapamil controlled release
- 2 (Active Comparator): 300 mg capsule of Verelan PM or 300 mg verapamil controlled release capsule given orally with food as a single dose with blood collected at 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 14, 16, 24, 30, 36, 48, 60 and 72 hours.
  Interventions: Drug: verapamil controlled release

INTERVENTIONS:
Drug: verapamil controlled release — verapamil 300 mg controlled release capsule as a single dose
  Other Names: Verelan PM; verapamil controlled release capsule

SUMMARY:
The purpose of this study is to determine the bioequivalency of Synerx Pharma Verapamil extended release capsules.

DETAILED DESCRIPTION:
The purpose of this study is to determine if Synerx Pharma Verapamil HCl ER Capsules are bioequivalent to Verelan PM capsules in healthy volunteers under food effect conditions.

ELIGIBILITY:
Inclusion Criteria:

Healthy adult male or female volunteers, 18-55 years of age. Subjects will be continuous non-smokers for at least 3 months prior to the first dose.

Weighing at least 60 kg for males and 52 kg for females and within the normal range according to accepted normal values of the Body Mass Index Chart (18.00 -28.00 kg/m2).

Medically healthy subjects with clinically normal laboratory profiles, vital signs and ECGs.

Absence of any exclusion criteria during history, physical, or laboratory evaluation.

Confirmation that all female subjects are not pregnant by a certified, validated pregnancy test.

Females of childbearing potential should either be sexually inactive (abstinent) for 14 days prior to the first dose and throughout the study or be an acceptable birth control method Postmenopausal women with amenorrhea for at least 2 years will be eligible. Give voluntary written informed consent to participate in the study.

Exclusion Criteria:

History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease.

In addition, history or presence of: alcoholism or drug abuse within the past year; hypersensitivity or idiosyncratic reaction to verapamil, other calcium ion influx inhibitors or any other component of the product formulations; idiosyncratic reaction to acetaminophen; malabsorption within the past year; recurrent headaches or migraines. Presence of a medical condition requiring regular treatment with prescription drugs.

Tests giving reasonable suspicion of a disease that would contraindicate taking an investigational drug or that might affect the interpretation of the results of the study.

Female subjects who are pregnant or lactating. Subjects who tested positive at screening for HIV, HbsAg or HCV. Positive test results for drugs of abuse or alcohol. Subjects whose sitting blood pressure is less than 110/60 mmHg at screening or 100/55 mmHg prior to dosing in each period.

Subjects whose pulse is lower than 55 b.p.m. at screening or 50 b.p.m. prior to dosing in each period.

Subjects whose PR interval is >190 msec at screening and >200 msec prior to dosing in each period.

Subjects whose QTc interval is >450 msec at screening and prior to dosing in each period.

Subjects who have used any drugs or substances known to be strong inducers and/or inhibitors of CYP enzymes within 28 days prior to the first dose.

Subjects who have been on a special diet during the 28 days prior to the first dose and throughout the study.

Subjects who donated 50 to 499 mL of blood within 30 days and more than 499 mL within 56 days prior to the first dose.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2007-07; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | 72 hours
  Statistical comparison of verapamil blood levels obtained over 72 hours when dosed with either the Verelan PM capsule or Synerx Pharma verapamil controlled release capsule. The comparison will compare Cmax and AUC and provide 80 to 125% confidence intervals for the values.

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Morelli, MD, Principal Investigator — MDS Pharma